CLINICAL TRIAL: NCT03713684
Title: A 56-week, Multicenter, Double-blind, Placebo-controlled, Randomized Study to Evaluate the Efficacy and Safety of Efpeglenatide Once Weekly in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Basal Insulin Alone or in Combination With Oral Antidiabetic Drug(s)
Brief Title: Efficacy and Safety of Efpeglenatide Versus Placebo in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Basal Insulin Alone or in Combination With Oral Antidiabetic Drug(s)
Acronym: AMPLITUDE-L
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to cancel TRIAL, not related to safety concern
Sponsor: Sanofi (Industry)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14893; U1111-1189-5009 (Other: UTN)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo (matched to efpeglenatide) subcutaneous (SC) injection once weekly up to Week 56 on top of basal insulin alone or in combination with oral antidiabetic drugs (OADs).
  Interventions: Drug: Placebo; Drug: Background therapy
- Efpeglenatide 2 mg (Experimental): Participants received Efpeglenatide 2 milligrams (mg) SC injection once weekly up to Week 56 on top of basal insulin alone or in combination with OADs.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy
- Efpeglenatide 4 mg (Experimental): Participants received Efpeglenatide 4 mg SC injection once weekly up to Week 56 on top of basal insulin alone or in combination with OADs. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg and maintained at the 4 mg dose through-out the treatment duration up to Week 56.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy
- Efpeglenatide 6 mg (Experimental): Participants received Efpeglenatide 6 mg SC injection once weekly up to Week 56 on top of basal insulin alone or in combination with OADs. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg until Week 4 and later up-titrated to 6 mg and maintained at the 6 mg dose through-out the treatment duration up to Week 56.
  Interventions: Drug: Efpeglenatide SAR439977; Drug: Background therapy

INTERVENTIONS:
Drug: Efpeglenatide SAR439977 — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Efpeglenatide 2 mg; Efpeglenatide 4 mg; Efpeglenatide 6 mg
Drug: Placebo — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Arms: Placebo
Drug: Background therapy — Lantus (Insulin Glargine), SC, once daily; OADs, administered as per investigator prescription and in accordance with local labeling.

SUMMARY:
Primary Objective:

To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo in glycated hemoglobin (HbA1c) change in participants with type 2 diabetes mellitus (T2DM) inadequately controlled with basal insulin alone or in combination with oral antidiabetic drugs (OADs).

Secondary Objectives:

* To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo on glycemic control.
* To demonstrate the superiority of once weekly injection of efpeglenatide in comparison to placebo on body weight.
* To evaluate the safety of once weekly injection of efpeglenatide.

DETAILED DESCRIPTION:
Study duration per participant was approximately 64 weeks including an up to 2-week Screening Period, a 30-week Core Treatment Period, a 26-week Safety Extension Period, and a 6-week safety Follow-up Period.

ELIGIBILITY:
Inclusion criteria:

* Participant must be greater than or equal to (>=)18 years of age at the time of signing the informed consent.
* Participants with T2DM.
* Diabetes diagnosed at least 1 year before screening.
* Participants on basal insulin regimen alone or in combination with OADs for at least 6 months prior to screening.
* HbA1c between 7.0 percent (%) and 10.0% (inclusive) measured by the central laboratory at screening.

Exclusion criteria:

* History of severe hypoglycemia requiring emergency room admission or hospitalization within 3 months prior to screening.
* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months prior to screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to) gastroparesis, unstable and not controlled gastroesophageal reflux disease requiring medical treatment within 6 months prior to screening.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy has been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (e.g., multiple endocrine neoplasia syndromes).
* Body weight change of >=5 kilograms within the last 3 months prior to screening.
* Systolic blood pressure greater than (>)180 millimetres of mercury (mmHg) and/or diastolic blood pressure >100 mmHg at randomization.
* End-stage renal disease as defined by estimated glomerular filtration rate (by Modification of Diet in Renal Disease) of less than 15 mL/min/1.73 m^2.
* Laboratory findings at the screening Visit:

  * Alanine aminotransferase or aspartate aminotransferase >3 * upper limit of normal (ULN) or total bilirubin >1.5*ULN (except in case of documented Gilbert's syndrome);
  * Amylase and/or lipase: >3*ULN;
  * Calcitonin >=5.9 picomoles per liter (pmol/L) (20 picograms per milliliter [pg/mL]).
* Gastric surgery or other gastric procedures intended for weight loss within 2 years prior to screening, or planned during study period.
* Pregnant (confirmed by serum pregnancy test at screening) or breast-feeding women.
* Women of childbearing potential not willing to use highly effective method(s) of birth control or who were unwilling to be tested for pregnancy during the study period and for at least 5 weeks after the last dose of study intervention.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- United States (22):
  - Investigational Site Number 8400038, Birmingham, Alabama
  - Investigational Site Number 8400035, Chandler, Arizona
  - Investigational Site Number 8400005, Glendale, Arizona
  - Investigational Site Number 8400057, Huntington Park, California
  - Investigational Site Number 8400058, La Jolla, California
  - Investigational Site Number 8400009, Los Angeles, California
  - Investigational Site Number 8400045, Spring Valley, California
  - Investigational Site Number 8400040, Tustin, California
  - Investigational Site Number 8400026, Van Nuys, California
  - Investigational Site Number 8400055, Orlando, Florida
  - Investigational Site Number 8400041, Pembroke Pines, Florida
  - Investigational Site Number 8400025, Lawrenceville, Georgia
  - Investigational Site Number 8400052, West Des Moines, Iowa
  - Investigational Site Number 8400044, Lexington, Kentucky
  - Investigational Site Number 8400001, Bridgeton, New Jersey
  - Investigational Site Number 8400039, New Windsor, New York
  - Investigational Site Number 8400036, Morehead City, North Carolina
  - Investigational Site Number 8400013, Maumee, Ohio
  - Investigational Site Number 8400030, Dallas, Texas
  - Investigational Site Number 8400063, Dallas, Texas
  - Investigational Site Number 8400043, San Antonio, Texas
  - Investigational Site Number 8400037, Layton, Utah
- China (9):
  - Investigational Site Number 1560005, Baotou
  - Investigational Site Number 1560017, Beijing
  - Investigational Site Number 1560006, Changsha
  - Investigational Site Number 1560001, Chengdu
  - Investigational Site Number 1560004, Shanghai
  - Investigational Site Number 1560036, Shanghai
  - Investigational Site Number 1560012, Shanghai
  - Investigational Site Number 1560013, Shanghai
  - Investigational Site Number 1560003, Zhengzhou
- South Korea (16):
  - Investigational Site Number 4100009, Busan
  - Investigational Site Number 4100001, Daejeon
  - Investigational Site Number 4100016, Gwangju
  - Investigational Site Number 4100010, Gwangju
  - Investigational Site Number 4100013, Gyeonggi-do
  - Investigational Site Number 4100015, Incheon
  - Investigational Site Number 4100014, Jeonju
  - Investigational Site Number 4100007, Seongnam-si
  - Investigational Site Number 4100008, Seoul
  - Investigational Site Number 4100002, Seoul
  - Investigational Site Number 4100005, Seoul
  - Investigational Site Number 4100004, Seoul
  - Investigational Site Number 4100003, Seoul
  - Investigational Site Number 4100011, Seoul
  - Investigational Site Number 4100006, Seoul
  - Investigational Site Number 4100012, Suwon

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) by SANOFI: Product rights transferred to Hanmi Pharmaceutical.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 47 active sites in 3 countries. A total of 540 participants were screened between 09 November 2018 and 02 September 2020, out of which 170 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 370 participants were randomized in 1:1:1:1 ratio to either placebo, efpeglenatide 2 milligrams (mg), efpeglenatide 4 mg, or efpeglenatide 6 mg treatment arms, stratified by screening glycated hemoglobin (HbA1c) values (less than [<]8%, greater than or equal to [>=]8%) and sulfonylurea (SU) use at screening (Yes/No).
Groups:
- Efpeglenatide 4 mg: Participants received Efpeglenatide 4 mg SC injection once weekly up to Week 56 or in combination with OADs. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg and maintained at the 4 mg dose through-out the treatment duration up to Week 56.
- Efpeglenatide 6 mg: Participants received Efpeglenatide 6 mg SC injection once weekly up to Week 56 or in combination with OADs. Participants initiated dosing at 2 mg once weekly up to Week 1; which was up titrated to 4 mg until Week 4 and later up-titrated to 6 mg and maintained at the 6 mg dose through-out the treatment duration up to Week 56.
Period: Overall Study
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Started | 92 | 92 | 93 | 93
Safety Population (Participants who received at least 1 dose or part of a dose of the Investigational Medicinal Product (IMP), analyzed according to the treatment actually received.) | 92 | 92 | 96 (For safety analysis participants were included in the treatment arm that they were exposed for longer duration. 3 participants randomized to Efpeglenatide 6 mg arm received 4 mg dose for longer duration; and considered in Efpeglenatide 4 mg arm for safety analysis.) | 90
Completed 30-Week Core Treatment Period | 50 | 52 | 51 | 49
Completed (Completed 56-Week treatment period.) | 6 | 5 | 5 | 6
Not Completed | 86 | 87 | 88 | 87
Not completed — Adverse Event | 1 | 3 | 1 | 0
Not completed — Poor compliance to protocol | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 14 | 6 | 14 | 16
Not completed — Other than specified | 69 | 77 | 73 | 70

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population which included all participants randomized irrespective of compliance with the study protocol and procedures analyzed, according to the treatment group allocated by randomization.
Groups:
- Placebo: Participants received placebo (matched to efpeglenatide) SC injection once weekly up to Week 56 on top of basal insulin alone or in combination with OADs.
- Efpeglenatide 2 mg: Participants received Efpeglenatide 2 mg SC injection once weekly up to Week 56 on top of basal insulin alone or in combination with OADs.
- Total: Total of all reporting groups
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Total
Number analyzed (Participants) | 92 | 92 | 93 | 93 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.7) | 59.1 (10.7) | 60.6 (11.5) | 61.6 (10.3) | 60.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 42 | 42 | 40 | 173
  Male | 43 | 50 | 51 | 53 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 49 | 51 | 50 | 195
  Black or African American | 9 | 9 | 10 | 8 | 36
  Asian | 36 | 33 | 30 | 34 | 133
  Other | 2 | 1 | 1 | 1 | 5
  Unknown | 0 | 0 | 1 | 0 | 1
Baseline Glycated Hemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.54 (0.83) | 8.42 (0.79) | 8.46 (0.79) | 8.40 (0.72) | 8.46 (0.78)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: Here, 'number analyzed' = participants with available data for the specified baseline measure.
  kilogram per square meter (kg/m^2)
    number analyzed (Participants) | 91 | 92 | 93 | 93 | 369
    (all) | 30.1 (5.6) | 31.1 (6.1) | 30.0 (6.6) | 31.0 (7.1) | 30.6 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 30 in HbA1c
Time Frame: Baseline to Week 30
Population: Analysis was performed on intent to treat (ITT) population which included all randomized participants, irrespective of compliance with the study protocol and procedures analyzed, according to the treatment group allocated by randomization. Here, "Overall number of participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 59 | 63 | 60 | 63
percentage of HbA1c | -0.33 (1.09) | -1.27 (0.95) | -1.24 (0.96) | -1.43 (0.94)

2. Secondary Outcome: Number of Participants With HbA1c <7.0% at Week 30
Description: Participants who had no available assessment for HbA1c at Week 30 were considered as non-responders.
Time Frame: Week 30
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 92 | 92 | 93 | 93
Participants | 10 | 32 | 28 | 40

3. Secondary Outcome: Change From Baseline to Week 56 in HbA1c
Description: This analysis included Week 56 assessment performed per protocol as well as premature end of treatment/study visit recorded as Week 56 due to early termination.
Time Frame: Baseline to Week 56
Population: Analysis was performed on ITT population. Here, "Overall number of participants analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 9 | 8 | 10 | 14
percentage of HbA1c | -0.32 (0.86) | -1.08 (0.77) | -1.23 (0.88) | -1.16 (1.34)

4. Secondary Outcome: Change From Baseline to Week 30 in Fasting Plasma Glucose (FPG)
Time Frame: Baseline to Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 54 | 55 | 51 | 56
millimoles per liter (mmol/L) | -0.41 (3.00) | -1.34 (2.80) | -1.33 (3.52) | -2.22 (1.89)

5. Secondary Outcome: Change From Baseline to Week 30 and Week 56 in Body Weight
Description: as for outcome 3
Time Frame: Baseline to Week 30 and Week 56
Population: Analysis was performed on ITT population. Here, "Overall number of participants analyzed"= participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified row.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 60 | 64 | 61 | 62
kilograms
  Week 30 | 0.29 (3.23) | -0.68 (3.63) | -1.99 (3.13) | -3.14 (3.19)
  Week 56: number analyzed (Participants) | 10 | 8 | 15 | 15
  Week 56 | 0.66 (3.22) | -2.39 (10.69) | -1.77 (5.36) | -2.85 (4.80)

6. Secondary Outcome: Number of Participants With At Least One Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL], and Severe Hypoglycemia)
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <54 mg/dL (<3.0 mmol/L). Severe hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline up to Week 56
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 92 | 92 | 96 | 90
Participants
  Documented symptomatic hypoglycemia (<54 mg/dL) | 4 | 8 | 10 | 9
  Severe hypoglycemia | 1 | 2 | 1 | 2

7. Secondary Outcome: Number of Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL] and Severe Hypoglycemia) Per Participant-Year
Description: as for outcome 6
Time Frame: Baseline up to Week 56
Population: Analysis was performed on safety population.
Measure: Number; unit: events per participant-year
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Number analyzed (Participants) | 92 | 92 | 96 | 90
events per participant-year
  Documented symptomatic hypoglycemia (<54 mg/dL) | 0.07 | 0.27 | 0.45 | 0.46
  Severe hypoglycemia | 0.09 | 0.05 | 0.05 | 0.04

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent up to end of study (up to Week 62). Time frame for reporting of treatment emergent adverse events (TEAEs) was from first injection of Investigational Medicinal Product (IMP) up to 30 days after the last injection of the IMP (i.e. up to Week 60).
Description: TEAEs were defined as AEs that developed or worsened, or became serious during the treatment-emergent period (time from first injection of IMP up to 30 days after the last injection of the IMP [i.e. up to Week 60]). Analysis was performed on safety population.
Arm/Group | Placebo | Efpeglenatide 2 mg | Efpeglenatide 4 mg | Efpeglenatide 6 mg
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92 | 0/96 | 0/90
Serious Adverse Events (participants affected / at risk) | 9/92 | 7/92 | 5/96 | 10/90
Other Adverse Events (participants affected / at risk) | 25/92 | 33/92 | 42/96 | 46/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | Efpeglenatide 2 mg (N=92) | Efpeglenatide 4 mg (N=96) | Efpeglenatide 6 mg (N=90)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Troponin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | Efpeglenatide 2 mg (N=92) | Efpeglenatide 4 mg (N=96) | Efpeglenatide 6 mg (N=90)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (9) | 4 (4) | 4 (6) | 5 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 11 (11) | 13 (14)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (6) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 5 (5) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 10 (15) | 15 (19) | 14 (19)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (17) | 19 (21) | 16 (24)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (5) | 12 (13) | 9 (13)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Amylase Increased (Investigations) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
Lipase Increased (Investigations) | 2 (2) | 9 (10) | 4 (4) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor on 09 September 2020. Due to early termination of the study, few efficacy evaluations originally planned in the protocol were no longer considered to be relevant and were not performed. Primary, and secondary efficacy data were descriptively summarized and data were carefully considered given that the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03713684/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03713684/SAP_001.pdf